CLINICAL TRIAL: NCT06252428
Title: Detection of Biofilm Among Uropathogenic Escherichia Coli Clinical Isolates in Suez Canal University Hospitals
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Other Study IDs: Moshera Ahmed Sherif Sherif
Record Dates: First submitted 2024-01-30; First posted 2024-02-09 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Escherichia Coli Infections
Keywords: Uropathogenic E. coli; biofilm; antibiotic resistance; MTCP; CRA
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine specimens will be collected under aseptic precautions from clinically suspected patients with UTIs in different wards in Suez Canal University hospitals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This descriptive cross-sectional study will beconducted in Suez Canal University Hospitals (SCUHs) in Ismailia, Egypt. The study aims to detect Escherichia coli biofilm producers to improve prognosis and treatment and reduce morbidity and mortality rates due to this infection.

DETAILED DESCRIPTION:
Forty seven clinical isolates of non-duplicated UPEC will be collected from clinically suspected cases of UTI in different departments in SCUHs. Isolates will be identified as E. coli by colony morphology, Gram staining and biochemical reactions. Antimicrobial sensitivity testing will be performed by Kirby-Bauer disc diffusion method on Muller-Hinton agar plate. The detection of biofilm will be carried out by Congo Red Agar (CRA) method and modified tissue culture plate (MTCP) method.

ELIGIBILITY:
Inclusion Criteria:

* Patients showing criteria for Symptomatic Urinary Tract Infection (SUTI) according to Center of Diseases and Control criteria (CDC) (CDC, 2022).

Patient has at least one of the following signs or symptoms:

* fever (>38.0°C)
* suprapubic tenderness
* costovertebral angle pain or tenderness
* urinary urgency
* urinary frequency
* dysuria

Exclusion Criteria:

* 1. Patients received antibiotic treatment in the last 48 hours 2. Refusal of the patients to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients of both sexes and all age groups attending different departments in Suez Canal University hospitals.
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
antibiotic resistance | from 18-24 hours
  Susceptibility testing will be performed according to the standard Kirby-Bauer disk diffusion method on Mueller Hinton agar and interpreted according to the Clinical and Laboratory Standard Institute (CLSI) guidelines. Antibiotic discs include Amoxicillin-clavulanate, Piperacillin-tazobactam, Cefotaxime, Ceftazidime, Aztreonam, Imipenem, Gentamicin, Amikacin, Norfloxacin, ciprofloxacin, levofloxacin, Trimethoprim-sulfamethoxazole, Nitrofurantoin.
Congo red Agar method (CRA) | 24 to 48 hours
  The medium will be prepared by adding 37 gm brain heart infusion (BHI) powder, 50 gm sucrose and 10 gm agar to 900 ml distilled water and autoclaved at 121°C for 15 minutes. Congo red will be prepared separately by dissolving 0.8 gm of congo red stain in 100 ml distilled water as concentrated aqueous solution and autoclaved at 121°C for 15 minutes and thenit will be added to the previous media when it cooled to 55°C. The congo red agar will be distributed in sterile plates. Plates will be inoculated by the test bacteria and incubated aerobically for 24 to 48 hours at 37°C. Positive results will be indicated by black colonies with a dry crystalline consistency. Weak slime producers usually remain pink.
Modified tissue culture plate method (MTCP) | up to 24 hours
  All isolates will be screened for their ability to form biofilm by the TCP method with a modification in duration of incubation, which will be extended to 24 hours and the addition of glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Rania Kishk, professor, Study Chair — Faculty of Medicine - Suez Canal University
Locations (1):
- Faculty of Medicine, Suez canal university, Ismailia, Egypt